CLINICAL TRIAL: NCT05188586
Title: New Onset Diabetes Management for Earlier Detection of Pancreatic Cancer (NODMED)
Acronym: NODMED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment targets not met
Sponsor: ClearNote Health (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: NODMED
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer
Keywords: Early Detection; New Onset Diabetes
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancreatic Cancer Signal Detection = Detected (Other): Subjects with test results "detected" will undergo MRI/Imaging
  Interventions: Other: MRI/Imaging
- Pancreatic Cancer Signal Detection = Not Detected (No Intervention)

INTERVENTIONS:
Other: MRI/Imaging — Blood collection and pancreatic cancer early detection testing with return of results.
  Arms: Pancreatic Cancer Signal Detection = Detected

SUMMARY:
Bluestar Genomics has developed a non-invasive test that aids in detection of occult pancreatic cancer in patients with new onset type II diabetes (NOD) who are 50 years old or older. The purpose of this study is to evaluate the performance of Bluestar Genomics early-detection pancreatic cancer test in a clinical setting. The study is prospective, longitudinal and interventional; tests will be ordered and results returned to site-investigators. If the test returns a pancreatic cancer signal "detected" result the study participant will undergo MRI imaging to evaluate for the presence of pancreatic cancer. The study is planned to enroll 6,550 newly diagnosed type 2 diabetic subjects according to inclusion and exclusion criteria.

DETAILED DESCRIPTION:
This is a prospective longitudinal and interventional study of the Bluestar Genomics early detection pancreatic cancer test. The test will be ordered and results returned to site-investigators. The study is planned to enroll 6,550 male and female, ≥ 50 years of age and newly diagnosed with type II diabetes (within 90 days prior to enrollment). NOD subjects will be assessed for eligibility and consented. Each subject can undergo up to 2 blood draws and electronic medical record search at 12 months from diabetes diagnosis.

The study population will be targeted to enroll a subjects with a BMI < 32. Subjects ≥ 50 years of age will be divided into two cohorts based on age as described below:

Cohort 1 = 65 years old or older Time 0 (T0) = blood draw within 90 days of diabetes diagnosis Time 1 (T1) = blood draw 6 month draw from diabetes diagnosis Time 2 (T2) = 12 months from diabetes diagnosis, no blood draw, only medical record search for all patients for evidence of pancreatic neoplasia developed after T1.

Cohort 2 = 50 - 64 years old Time 0 (T0) = blood draw within 90 days of diabetes diagnosis Time 1 (T1) = blood draw 6 month draw from diabetes diagnosis Time 2 (T2) = 12 months from diabetes diagnosis, no blood draw, only medical record search for all patients for evidence of pancreatic neoplasia developed after T1.

Imaging Strategy MRI imaging (or alternate imaging if subject is unable to undergo MRI) will be performed on subjects whose test result is "detected".

If the imaging study results are abnormal, the subject will be referred back to their enrolling clinician for additional diagnostic work up as part of routine healthcare. If pancreatic cancer or other pancreatic lesion is diagnosed, the diagnostic reports will be collected as part of the study clinical data.

ELIGIBILITY:
Inclusion Criteria:

≥ 50 years of age or older at the time of enrollment

Willing to sign the informed consent form

Must have 2 occurrences from among the below parameters of diabetes mellitus (PDMs) in past 90 days measured in outpatient setting (not in urgent care, emergency room or while inpatient):

FBG ≥126mg/dl HbA1c ≥6.5% RBG ≥ 200mg/dl 2-hour post-glucose ≥200mg/dl (OGTT)

Must have had glycemic parameter measured in 3-18 months prior to screening that did NOT meet DM criteria

Must be willing to provide several tubes of blood without endangering health

No history of pancreatic cancer or other known pancreatic neoplasia

No active cancers within the past 5 years (with the exception of non-melanoma skin cancers resolved/treated > 1 year prior to enrollment and in situ cancers)

Exclusion Criteria:

Prior DM diagnosis

Met criteria for DM ≥91 days prior to enrollment (patients with prior gestational diabetes that has resolved are NOT acceptable to enroll)

Carried a DM diagnosis or used anti-DM medications at a time greater than or equal to 91 days prior to enrollment

Any known pancreatic lesions (aside from diabetes)

Received cancer treatment within the past 5 years (with the exception of treatment of non-melanoma skin cancer), carrying a current cancer diagnosis, and/or being investigated for suspicion of past cancer recurrence.

Current chronic or acute oral steroid use

History of intra-articular steroid injections (<1 week) of the qualifying DM blood test (allowed exception: nasal, topical, oral budesonide)

Any surgery requiring general anesthesia within 2 months of collection

Local anesthetic (including dental novocaine) within 1 week of collection

History or presence of HIV/AIDs, Hepatitis A or E within the past five years, TB, any kind of prion disorder (e.g., CJD)

Blood transfusion within 1 month

Organ transplant recipient

Currently pregnant, or pregnancy within last 12 months

Receipt of systemic immunomodulation therapy within past 12 months

Significant medical condition that in the site investigator's opinion would compromise the subject's ability to tolerate study interventions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) | 12 months or until diagnostic resolution
  defined as the proportion of participants with pancreatic neoplasia diagnosis out of all subjects with pancreatic signal "detected" test result.
Negative Predictive Value (NPV) | 12 months or until diagnostic resolution
  defined as the proportion of participants with no pancreatic neoplasia diagnosis out of all the subjects with pancreatic signal "not detected" test results.
Specificity | 12 months or until diagnostic resolution
  defined as the proportion of participants with pancreatic signal "not detected" results out of all subjects with no pancreatic neoplasia diagnosis.

SECONDARY OUTCOMES:
Time to pancreatic cancer diagnosis | 12 months or until diagnostic resolution
  Median time to pancreatic cancer diagnosis (using Pancreatic Cancer Signal Detection testing) relative to new onset diabetes (NOD) diagnosis compared to Median time to pancreatic cancer diagnosis relative to NOD diagnosis in the absence of Pancreatic Cancer Signal Detection testing, based on published data
Stage Shift | 12 months or until diagnostic resolution
  Stage Shift in NODs with Pancreatic Cancer in subjects that have undergone Pancreatic Cancer Signal Detection testing vs subjects without Pancreatic Cancer Signal Detection testing

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Levy, PhD, Principal Investigator — ClearNote Health
Locations (5):
- United States (5):
  - Headlands Research - Scottsdale - PPDS, Scottsdale, Arizona
  - JEM Research Institute - Headlands - PPDS, Atlantis, Florida
  - Prisma Health/Endocrinology specialist and Thyroid, Greenville, South Carolina
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Manassas Clinical Research Center, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: No